CLINICAL TRIAL: NCT06487091
Title: Analysis of Platelet Function During Impella Support
Brief Title: Platelet Function and Impella Support
Acronym: IMPELLA-PLT
Status: Recruiting | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: Abiomed Inc. (Industry)
Responsible Party: Principal Investigator, Filippo Consolo, Assistant Professor, IRCCS Ospedale San Raffaele
Other Study IDs: IMPELLA-PLT
Record Dates: First submitted 2024-05-31; First posted 2024-07-05 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Cardiogenic Shock; Cardiac Arrest; Mechanical Circulatory Support
Keywords: Cardiogenic Shock; Cardiac Arrest; Mechanical Circulatory Support; Impella; Platelet Function; Bleeding; Thrombosis; Hemolyisis; platelet microRNA
MeSH Terms: conditions — Shock, Cardiogenic; Heart Arrest; Hemorrhage; Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- patients on Impella support: CS/CA patients that receive primary temporary mechanical circulatory support with an Impella device
  Interventions: Diagnostic Test: Analysis of platelet function

INTERVENTIONS:
Diagnostic Test: Analysis of platelet function — Blood withdrawal, platelet separation and analysis of the expression levels of markers of platelet function

SUMMARY:
Mechanical circulatory support (MCS) with the Impella microaxial pump in the setting of cardiogenic shock/cardiac arrest (CS/CA) is accompanied by substantial risk of life-threatening complications, including hemolysis, thrombotic and bleeding events.

Previous studies in patients on durable MCS suggest that device-induced platelet dysfunction plays a major contributory role in the development of such events and that selected markers of platelet function have the potential to stratify patients according to an elevated risk of adverse events. To date, the potential clinical utility of markers of altered platelet function in patients supported with an Impella pump is unexplored.

The proposed study will analyze changes in platelet function in the setting of Impella support (primary aim) and possibly identify a platelet function "profile" indicative of patients at high-risk to develop adverse events (secondary aim).

The study is a prospective observational study. Changes in the expression levels of markers of both platelet activation and aggregation in patients supported with an Impella pump will be measured. Data will be longitudinally measured: pre-implant (before Impella implantation) and then after 24, 48 and 72h of Impella support. Markers that will be analyzed include surface platelet receptors and platelet microRNAs. Experimental data will be correlated with clinical outcomes, including the occurrence of adverse events.

This study will provide mechanistic insights into the effect of Impella support on the protein and miRNA expression of platelets. The intention is to get a better understanding of distinct pathways of platelet function related to Impella support and their relationship to adverse events. Our data might open the perspective for the future clinical use of markers of platelet function to enhance the early recognition of patients at high risk of developing an adverse event and the definition of novel, personalized therapeutic strategies targeted to platelet biology to prevent their occurrence.

DETAILED DESCRIPTION:
STUDY DESIGN AND MAIN OBJECTIVE Prospective observational study to evaluate changes in the expression levels of markers of platelet function (activation and aggregation capacity) in CS/CA patients who receive an Impella device for temporary mechanical circulatory support

HYPOTHESIS

* progressive change of platelet function occurs over the course of Impella support driven by shear forces exerted by the pump on recirculating blood
* markers of changes in platelet function can be identified at the protein and nuclear level in platelet samples extracted form patients supported with an Impella pump
* specific trends of the changes of the expression levels of markers of platelet function might allow identifying patients at higher risk of developing a thrombotic/hemorrhagic complication
* the expression levels of markers of platelet function are indeed altered in patients even before the clinical manifestation of the event

METHODOLOGY The markers that will be analyzed have been selected according to recent studies showing

* significant changes in their expression levels driven by durable MCS devices
* their potential to identify patients at high risk of developing adverse events
* their association with coagulation/hemostatic disorders and hemolysis and include:
* platelet receptors GPIba, GPIIb/IIIa, and GPVI [1-4].
* platelet microRNA miR-20b-5p, miR-25-3p, miR-126-5p, miR-451a, miR-320a, miR-223-3p, miR-144-rp, miR-151a-3p, and miR-454-3p [5]. The expression levels of these microRNAs will be measured in both PRP and PPP samples, to confirm their actual expression by platelets.

Data will be measured

* pre-implant (i.e., immediately prior to Impella implantation), to evaluate the patient-specific baseline profile, and then following
* 24 hours, 48 hours, and 72 hours of Impella support. This way it will possible to quantify longitudinal changes in the levels of expression of the selected markers over the course of Impella support (vs. baseline).

Data will be also measured during the acute phase of any of the following adverse events that will occur during Impella support (not limited to 72 hours):

* thrombosis (of the patient - any site - and of the pump)
* ischemic/hemorrhagic stroke
* any surgical or non-surgical bleeding
* hemolysis Adverse events will be defined according to most recent criteria [6-8].

Furthermore, inferences of any change in the anticaogulation regimen that may occur over the course of Impella support (not limited to 72 hours) will be evaluated: to this aim, markers of platelet function will be analyzed 12 hours following any change in the anticoagulation regimen.

Experimental data will be correlated with clinical outcomes, including the occurrence of adverse events, to possibly identify an "event-related platelet function profile" characteristics of the sub-group of patients that will develop adverse events. The occurrence of adverse events will be continuously recorded over the whole duration of Impella support.

TREATMENT PROCEDURE To measure the expression levels of the selected markers of platelet function, platelet samples will be isolated from patients' blood (10-mL volume) via standard laboratory techniques. The expression levels of the analyzed markers will be measured via quantitative real-time polymerase chain reaction and protein quantitation/function assay, such as enzyme-linked immunosorbent assay.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18yrs-old and <75yrs-old
* Cardiogenic shock SCAI class C-D-E
* primary tMCS with an Impella device (all Impella pumps)
* Informed consent

Exclusion Criteria:

* Patients <18yrs-old or >75yrs-old
* Refusal to participate to the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CS/CA patients who receive temporary mechanical circulatory support with an Impella device
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-01-24 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Expression levels of platelet surface markers of activation and aggregation and platelet microRNAs in patients on Impella support | baseline (prior to Impella implantation) vs. 24 hours, 48 hours and 72 hours of Impella support
  Changes (measured as percentage variation) in the expression levels of platelet surface markers of activation and aggregation (GPIba, GPIIb/IIIa, and GPVI) and platelet microRNA (miR-20b-5p, miR-25-3p, miR-126-5p, miR-451a, miR-320a, miR-223-3p, miR-144-rp, miR-151a-3p, and miR-454-3p) during tMCS with an Impella device (all Impella pumps)

SECONDARY OUTCOMES:
Expression levels of platelet surface markers of activation and aggregation and platelet microRNAs in the acute phase of an adverse event (hemolysis, thrombosis, bleeding). Adverse events will be determined according to [6-8] | immediately after any adverse event, anticipated average 30 days
  Expression levels of platelet surface markers of activation and aggregation (GPIba, GPIIb/IIIa, and GPVI) and platelet microRNA (miR-20b-5p, miR-25-3p, miR-126-5p, miR-451a, miR-320a, miR-223-3p, miR-144-rp, miR-151a-3p, and miR-454-3p) measured following the occurrence of an adverse event (hemolysis, thrombosis, bleeding)
Expression levels of platelet surface markers of activation and aggregation and platelet microRNAs after any change in the antithrombotic regimen | 12 hours after any change in the antithrombotic regimen
  Expression levels of platelet surface markers of activation and aggregation (GPIba, GPIIb/IIIa, and GPVI) and platelet microRNA (miR-20b-5p, miR-25-3p, miR-126-5p, miR-451a, miR-320a, miR-223-3p, miR-144-rp, miR-151a-3p, and miR-454-3p) measured following any change in the antithrombotic regimen (lower dose and/or withdrawal of anticoagulant/antiplatelet drugs)

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Consolo, PhD, Study Chair — Università Vita-Salute San Raffaele; Mara Scandroglio, MD, Principal Investigator — Ospedale San Raffaele
Locations (2):
- Italy (2):
  - IRCCS San Raffaele Hospital, Milan
  - Università Vita Salute San Raffaele, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen Z, Mondal NK, Ding J, Gao J, Griffith BP, Wu ZJ. Shear-induced platelet receptor shedding by non-physiological high shear stress with short exposure time: glycoprotein Ibalpha and glycoprotein VI. Thromb Res. 2015 Apr;135(4):692-8. doi: 10.1016/j.thromres.2015.01.030. Epub 2015 Feb 7. PMID 25677981
- [Background] Klaeske K, Dieterlen MT, Eifert S, Scholz U, Garbade J, Jawad K, Sieg F, Borger MA, Meyer AL. Device-induced platelet dysfunction in patients after left ventricular assist device implantation. J Thromb Haemost. 2021 May;19(5):1331-1341. doi: 10.1111/jth.15279. Epub 2021 Mar 28. PMID 33636040
- [Background] Arias K, Sun W, Wang S, Sorensen EN, Feller E, Kaczorowski D, Griffith B, Wu ZJ. Acquired platelet defects are responsible for nonsurgical bleeding in left ventricular assist device recipients. Artif Organs. 2022 Nov;46(11):2244-2256. doi: 10.1111/aor.14319. Epub 2022 May 30. PMID 35596611
- [Background] Klaeske K, Meyer AL, Saeed D, Eifert S, Jawad K, Sieg F, Haunschild J, Borger MA, Dieterlen MT. Decreased Platelet Specific Receptor Expression of P-Selectin and GPIIb/IIIa Predict Future Non-Surgical Bleeding in Patients after Left Ventricular Assist Device Implantation. Int J Mol Sci. 2022 Sep 6;23(18):10252. doi: 10.3390/ijms231810252. PMID 36142161
- [Background] Lombardi M, Bonora M, Baldetti L, Pieri M, Scandroglio AM, Landoni G, Zangrillo A, Foglieni C, Consolo F. Left ventricular assist devices promote changes in the expression levels of platelet microRNAs. Front Cardiovasc Med. 2023 Jun 15;10:1178556. doi: 10.3389/fcvm.2023.1178556. eCollection 2023. PMID 37396581
- [Background] Bernhardt AM, Copeland H, Deswal A, Gluck J, Givertz MM; Chairs:; Co-Chairs:; Contributing Writers:; Chair:; Co-Chair:; Contributing Writers:; Chair:; Co-Chairs:; Contributing Writers:; Chair:; Co-Chair:; Contributing Writers:. The International Society for Heart and Lung Transplantation/Heart Failure Society of America Guideline on Acute Mechanical Circulatory Support. J Heart Lung Transplant. 2023 Apr;42(4):e1-e64. doi: 10.1016/j.healun.2022.10.028. Epub 2023 Feb 6. No abstract available. PMID 36805198
- [Background] Garcia-Garcia HM, McFadden EP, Farb A, Mehran R, Stone GW, Spertus J, Onuma Y, Morel MA, van Es GA, Zuckerman B, Fearon WF, Taggart D, Kappetein AP, Krucoff MW, Vranckx P, Windecker S, Cutlip D, Serruys PW; Academic Research Consortium. Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document. Circulation. 2018 Jun 12;137(24):2635-2650. doi: 10.1161/CIRCULATIONAHA.117.029289. PMID 29891620
- [Background] Kormos RL, Antonides CFJ, Goldstein DJ, Cowger JA, Starling RC, Kirklin JK, Rame JE, Rosenthal D, Mooney ML, Caliskan K, Messe SR, Teuteberg JJ, Mohacsi P, Slaughter MS, Potapov EV, Rao V, Schima H, Stehlik J, Joseph S, Koenig SC, Pagani FD. Updated definitions of adverse events for trials and registries of mechanical circulatory support: A consensus statement of the mechanical circulatory support academic research consortium. J Heart Lung Transplant. 2020 Aug;39(8):735-750. doi: 10.1016/j.healun.2020.03.010. Epub 2020 Apr 18. No abstract available. PMID 32386998